CLINICAL TRIAL: NCT00269451
Title: Assessing PTSD After Earthquake in Turkey
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Sheba Medical Center (Other Government)
Other Study IDs: PTSD Turkey
Record Dates: First submitted 2005-12-22; First posted 2005-12-23 (Estimated); Last update posted 2005-12-23 (Estimated); Status verified 2005-12

CONDITIONS: Post-Traumatic Stress Disorder
MeSH Terms: conditions — Stress Disorders, Post-Traumatic

STUDY DESIGN:
Observational Model: Defined Population | Time Perspective: Prospective

SUMMARY:
Assessing the prevalence and natural course of PTSD after the 1999 Turkish earthquake

ELIGIBILITY:
Inclusion Criteria:

* People were in the earthquake area while it occured

Exclusion Criteria:

* People were not in the earthquake area while it occured

Min Age: 0 Years | Sex: All
Age Groups: Child, Adult, Older Adult

CONTACTS AND LOCATIONS:
Overall Officials: Joseph Zohar, MD, Principal Investigator — Tel Aviv University